CLINICAL TRIAL: NCT01941095
Title: Multicenter, Open Label, Phase IIIb Study to Evaluate the Safety and Tolerability of Subcutaneous Tocilizumab as Monotherapy and/or in Combination With Methotrexate or Other Non-Biologic Disease-Modifying Antirheumatic Drugs in Patients With Rheumatoid Arthritis
Brief Title: A Study of Subcutaneous Tocilizumab as Monotherapy and/or in Combination With Non-Biologic Disease Modifying Anti-Rheumatic Drugs (DMARDs) in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28695; 2013-000359-42 (EudraCT Number)
Record Dates: First submitted 2013-08-30; First posted 2013-09-13 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Azathioprine; Chloroquine; Hydroxychloroquine; Leflunomide; Methotrexate; Sulfasalazine; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab 162 milligrams (mg) SC injection once a week (QW) either as monotherapy or in combination with methotrexate or other non-biologic DMARDs during the treatment period of 52 weeks. The choice of monotherapy or combination treatment is according to the physician's judgment up to Week 24. Depending upon the participant's response to study regimen at Week 24, participant may either continue/discontinue/switch to tocilizumab monotherapy or may lead to intensification of methotrexate/non-biologic DMARDs with tocilizumab at a fixed dose of 162 mg SC QW till Week 52. After Week 52, participants who remain in study will enter a 8 week wash-out period and then (from Week 60) will proceed to the extension phase until tocilizumab is commercially available in Greece. Permitted DMARDs include methotrexate, azathioprine, chloroquine, hydroxychloroquine, leflunomide, and sulfasalazine.
  Interventions: Drug: Azathioprine; Drug: Chloroquine; Drug: Hydroxychloroquine; Drug: Leflunomide; Drug: Methotrexate; Drug: Sulfasalazine; Drug: Tocilizumab

INTERVENTIONS:
Drug: Azathioprine — Participants may receive azathioprine as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Chloroquine — Participants may receive chloroquine as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Hydroxychloroquine — Participants may receive hydroxychloroquine as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Leflunomide — Participants may receive leflunomide as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Methotrexate — Participants may receive methotrexate as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Sulfasalazine — Participants may receive sulfasalazine as a concomitant therapy with tocilizumab as per physician's judgment at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Tocilizumab — Participants will receive tocilizumab at a fixed dose of 162 mg SC QW either as monotherapy or in combination with non-biologic DMARDs.
  Other Names: RoActemra, Actemra

SUMMARY:
This Phase IIIb, multicenter, open label, single arm study will evaluate the safety and efficacy of subcutaneous (SC) tocilizumab as monotherapy or in combination with methotrexate or other non-biologic DMARDs in participants with active rheumatoid arthritis who are either naïve to or have an inadequate response to prior non-biologic or/and biologic DMARDs. The anticipated time on study treatment is 52 weeks. Those participants who will complete the 60-week study period and have achieved Disease Activity Score 28 (DAS28) remission or a good European League Against Rheumatism (EULAR) response at 52 weeks will be eligible to enter the extension phase until tocilizumab is commercially available and reimbursed in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active rheumatoid arthritis according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria
* Oral corticosteroids (less than or equal to [</=] 10 milligrams per day [mg/day] prednisolone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs; up to the maximum recommended dose) are permitted if on a stable dose regimen for greater than or equal to [>/=] 4 weeks prior to baseline
* Permitted non biologic DMARDs are allowed if a stable dose for at least 4 weeks prior to baseline
* Receiving treatment on an outpatient basis, not including tocilizumab
* Females of childbearing potential and males with female partners of childbearing potential must agree to use a reliable means of contraception during the study; females of childbearing potential must use a reliable means of contraception for at least 3 month following the last dose of tocilizumab

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline
* Rheumatic autoimmune disease other than rheumatoid arthritis; secondary Sjögren's syndrome with rheumatoid arthritis is permitted
* Functional Class 4 as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile rheumatoid arthritis and/or rheumatoid arthritis before the age of 16
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Participants with lack of peripheral venous access
* Exposure to tocilizumab (either intravenous [IV] or SC) at any time prior to baseline
* Treatment with any investigational agent within 4 weeks (or five half-lives of the investigational drug, whichever is longer) of screening
* Previous treatment with any cell-depending therapies
* Treatment with IV gamma globulin, plasmapheresis within 6 months of baseline
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine (including uncontrolled diabetes mellitus), or gastrointestinal disease
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections
* Any major episode of infection requiring hospitalization of treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years
* Positive for hepatitis B surface antigen or hepatitis C antibody
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (except for basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years
* Pregnant or breast feeding women
* History of alcohol, drug or chemical abuse within 1 year prior to screening
* Neuropathies or other conditions that interfere with pain evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Greece (10):
  - District Gen. Hosp. of Athens Laiko; A Propedeutic Internal Medicine Clinic & Research Center, Athens
  - Laiko General Hospital; Dept. of Pathophysiology-Uni of Athens, Athens
  - Hippokratio Hospital; 2Nd Internal Medicine, Athens
  - ATTIKO Hospital_4th University Internal Medicine Clinic, Haidari
  - Uni General Hospital of Heraklion; Medicine and Rheumatology Clinical Immunology and Allergy Dept, Heraklion
  - Uni Hospital of Ioannina; Rheumatology, Ioannina
  - University General Hospital of Larissa; Rheumatology Unit, Larissa
  - University Hospital of Patras; Rheumatology, Pátrai
  - EUROMEDICA Geniki Kliniki Thessalonikis; Rheumatology Department, Thessaloniki
  - General Hospital of Thessaloniki HIPPOKRATIO; Clinical Immunology Unit,2nd Dept of Internal Medicine, Thessaloniki

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 9 locations in Greece
Pre-assignment Details: A total of 100 participants were enrolled, out of which 97 participants received treatment. Analyses were performed in 97 participants.
Groups:
- Tocilizumab: Participants received tocilizumab 162 milligrams (mg) subcutaneous (SC) injection once a week (QW) either as monotherapy or in combination with methotrexate or other non-biologic disease modifying anti-rheumatic drugs (DMARDs) during the treatment period of 52 weeks. The choice of monotherapy or combination treatment was according to the physician's judgment up to Week 24. Depending upon the participant's response to study regimen at Week 24, participant might either continue/discontinue/switch to tocilizumab monotherapy or may lead to intensification of methotrexate/non-biologic DMARDs with tocilizumab at a fixed dose of 162 mg SC QW till Week 52.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 97
Completed | 41
Not Completed | 56
Not completed — Insufficient therapeutic response | 13
Not completed — Anaphylaxis or serious hypersensitivity | 2
Not completed — Adverse Event | 11
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set included all recruited participants who received at least one dose of SC tocilizumab.
Groups:
- Tocilizumab: Participants received tocilizumab 162 mg SC injection QW either as monotherapy or in combination with methotrexate or other non-biologic DMARDs during the treatment period of 52 weeks. The choice of monotherapy or combination treatment was according to the physician's judgment up to Week 24. Depending upon the participant's response to study regimen at Week 24, participant might either continue/discontinue/switch to tocilizumab monotherapy or may lead to intensification of methotrexate/non-biologic DMARDs with tocilizumab at a fixed dose of 162 mg SC QW till Week 52.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.27 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score Based on 28 Joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR) Remission at Week 24
Description: DAS28-ESR score is a measure of participant's disease activity calculated using tender joint count in 28 joints (TJC28), swollen joint count in 28 joints (SJC28), patient global assessment of disease activity (PGA) (general health [GH]) using visual analog scale (VAS): 0 millimeter (mm)=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS, and acute phase response (ESR in millimeters per hour [mm/hr]). The score is calculated using the following formula: DAS28-ESR = [0.56 multiplied by (*) square root (√) of TJC28] plus (+) [0.28*√SJC28]+[0.70*the natural logarithm (ln) ESR]+[0.014*GH]. DAS28-ESR score varies from 0 to 10, where higher scores represent greater disease activity. DAS28-ESR score of less than (<) 2.6 represents DAS28-ESR remission.
Time Frame: Week 24
Population: Full analysis set. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants | 40

2. Secondary Outcome: Percentage of Participants Who Maintained DAS28-ESR Remission From Week 24 up to Week 52 Among Participants on Tocilizumab Monotherapy Since Week 24
Description: DAS28-ESR score is a measure of participant's disease activity calculated using TJC28, SJC28, PGA using VAS 0 mm=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS, and acute phase response (ESR in mm/hr) for a total possible score of 0 to 10. The score is calculated using the following formula: DAS28-ESR = [0.56 * √TJC28 + [0.28*√SJC28]+[0.70*ln ESR]+[0.014*GH]. DAS28-ESR score varies from 0 to 10, where higher scores represent greater disease activity. DAS28-ESR score <2.6 represents DAS28-ESR remission. The percentage reported for Week 24 is based on confirmation on switching to SC tocilizumab monotherapy.
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52
Population: Per protocol analysis. Overall number of participants analyzed = participants evaluable for this outcome measure. Here, Number analyzed = number of participants analyzed for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 80
percentage of participants
  Week 24 | 38.7
  Week 28: number analyzed (Participants) | 79
  Week 28 | 34.2
  Week 32: number analyzed (Participants) | 74
  Week 32 | 36.5
  Week 36: number analyzed (Participants) | 74
  Week 36 | 36.5
  Week 40: number analyzed (Participants) | 74
  Week 40 | 36.5
  Week 44: number analyzed (Participants) | 71
  Week 44 | 35.2
  Week 48: number analyzed (Participants) | 70
  Week 48 | 35.7
  Week 52: number analyzed (Participants) | 67
  Week 52 | 38.8

3. Secondary Outcome: Percentage of Participants Who Achieved DAS28-ESR Remission/Low Disease Activity (LDA) From Week 28 up to Week 52 Among Participants With Intensification of Methotrexate/Other Non-Biologic DMARDs in Combination With Tocilizumab Since Week 24
Description: DAS28-ESR score is a measure of participant's disease activity calculated using TJC28, SJC28, PGA using VAS 0 mm=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS, and acute phase response (ESR in mm/hr) for a total possible score of 0 to 10. The score is calculated using the following formula: DAS28-ESR = [0.56 * √TJC28 + [0.28*√SJC28]+[0.70*ln ESR]+[0.014*GH]. DAS28-ESR score varies from 0 to 10, where higher scores represent greater disease activity. DAS28-ESR score <2.6 represents DAS28-ESR remission. DAS28-ESR score greater than or equal to (>/=) 2.6 and <3.2 represents LDA.
Time Frame: Weeks 28, 32, 36, 40, 44, 48, 52
Population: Full analysis set. Overall number of participants analyzed = participants evaluable for this outcome measure. Here, Number analyzed = number of participants analyzed for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
percentage of participants
  Week 28: Remission | 5.1
  Week 32: Remission: number analyzed (Participants) | 74
  Week 32: Remission | 8.1
  Week 36: Remission: number analyzed (Participants) | 74
  Week 36: Remission | 4.1
  Week 40: Remission: number analyzed (Participants) | 74
  Week 40: Remission | 9.5
  Week 44: Remission: number analyzed (Participants) | 72
  Week 44: Remission | 6.9
  Week 48: Remission: number analyzed (Participants) | 71
  Week 48: Remission | 8.5
  Week 52: Remission: number analyzed (Participants) | 67
  Week 52: Remission | 6
  Week 28: LDA | 7.6
  Week 32: LDA: number analyzed (Participants) | 74
  Week 32: LDA | 1.4
  Week 36: LDA: number analyzed (Participants) | 74
  Week 36: LDA | 6.8
  Week 40: LDA: number analyzed (Participants) | 74
  Week 40: LDA | 6.8
  Week 44: LDA: number analyzed (Participants) | 72
  Week 44: LDA | 6.9
  Week 48: LDA: number analyzed (Participants) | 71
  Week 48: LDA | 4.2
  Week 52: LDA: number analyzed (Participants) | 67
  Week 52: LDA | 9

4. Secondary Outcome: Change From Baseline in DAS28-ESR up to Week 52
Description: DAS28-ESR score is a measure of participant's disease activity calculated using TJC28, SJC28, PGA using VAS 0 mm=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS, and acute phase response (ESR in mm/hr) for a total possible score of 0 to 10. The score is calculated using the following formula: DAS28-ESR = [0.56 * √TJC28 + [0.28*√SJC28]+[0.70*ln ESR]+[0.014*GH]. DAS28-ESR score varies from 0 to 10, where higher scores represent greater disease activity. A negative change from baseline indicates an improvement.
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
units on a scale
  Change at Week 2 | -0.99 [-1.33 to -0.64]
  Change at Week 4: number analyzed (Participants) | 95
  Change at Week 4 | -1.70 [-2.06 to -1.36]
  Change at Week 8: number analyzed (Participants) | 93
  Change at Week 8 | -2.20 [-2.54 to -1.84]
  Change at Week 12: number analyzed (Participants) | 87
  Change at Week 12 | -2.56 [-2.91 to -2.20]
  Change at Week 16: number analyzed (Participants) | 85
  Change at Week 16 | -2.59 [-2.91 to -2.27]
  Change at Week 20: number analyzed (Participants) | 82
  Change at Week 20 | -2.93 [-3.24 to -2.62]
  Change at Week 24: number analyzed (Participants) | 80
  Change at Week 24 | -3.14 [-3.45 to -2.83]
  Change at Week 28: number analyzed (Participants) | 79
  Change at Week 28 | -3.22 [-3.53 to -2.90]
  Change at Week 32: number analyzed (Participants) | 74
  Change at Week 32 | -3.34 [-3.66 to -3.01]
  Change at Week 36: number analyzed (Participants) | 74
  Change at Week 36 | -3.32 [-3.64 to -3.00]
  Change at Week 40: number analyzed (Participants) | 74
  Change at Week 40 | -3.40 [-3.73 to -3.07]
  Change at Week 44: number analyzed (Participants) | 71
  Change at Week 44 | -3.45 [-3.78 to -3.11]
  Change at Week 48: number analyzed (Participants) | 70
  Change at Week 48 | -3.42 [-3.76 to -3.08]
  Change at Week 52: number analyzed (Participants) | 67
  Change at Week 52 | -3.40 [-3.73 to -3.07]

5. Secondary Outcome: Number of Participants With American College of Rheumatology 20 (ACR20) Response
Description: ACR20 response was defined as >/=20% improvement from baseline in both TJC28 and SJC28 as well as in 3 out of 5 additional parameters: Separate patient and physician's global assessment of disease activity on VAS (0 mm=no disease activity to 100 mm=maximum disease activity, displayed on the 100 mm horizontal VAS), patient's assessment of pain on VAS (0 mm=no pain to 100 mm=unbearable pain, displayed on the 100 mm horizontal VAS), Health Assessment Questionnaire - Disability Index (HAQ-DI) (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without any difficulty to 3=unable to do), and acute phase response (ESR in mm/hr, for a total possible score of 0 to 10).
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
participants
  Week 2 | 19
  Week 4: number analyzed (Participants) | 95
  Week 4 | 19
  Week 8: number analyzed (Participants) | 93
  Week 8 | 23
  Week 12: number analyzed (Participants) | 87
  Week 12 | 9
  Week 16: number analyzed (Participants) | 85
  Week 16 | 13
  Week 20: number analyzed (Participants) | 82
  Week 20 | 16
  Week 24: number analyzed (Participants) | 80
  Week 24 | 9
  Week 28: number analyzed (Participants) | 79
  Week 28 | 13
  Week 32: number analyzed (Participants) | 74
  Week 32 | 10
  Week 36: number analyzed (Participants) | 74
  Week 36 | 11
  Week 40: number analyzed (Participants) | 74
  Week 40 | 10
  Week 44: number analyzed (Participants) | 72
  Week 44 | 12
  Week 48: number analyzed (Participants) | 71
  Week 48 | 13
  Week 52: number analyzed (Participants) | 67
  Week 52 | 15

6. Secondary Outcome: Percentage of Participants With Good, Moderate, or No Response According to European League Against Rheumatism (EULAR) Response Criteria
Description: Response to treatment was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 reduction from the baseline visit. Participants with a score lesser than or equal to (</=) 3.2 and reduction of greater than (>) 1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score </=5.1 with reduction of >0.6 to </=1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to </=1.2 points, or any score with reduction </=0.6 points, were assessed as having 'no response'.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
percentage of participants
  Week 2: Good response | 9.4
  Week 2: Moderate response | 44.8
  Week 2: No response | 45.8
  Week 4: Good response: number analyzed (Participants) | 95
  Week 4: Good response | 9.5
  Week 4: Moderate response: number analyzed (Participants) | 95
  Week 4: Moderate response | 38.9
  Week 4: No response: number analyzed (Participants) | 95
  Week 4: No response | 51.6
  Week 8: Good response: number analyzed (Participants) | 93
  Week 8: Good response | 10.8
  Week 8: Moderate response: number analyzed (Participants) | 93
  Week 8: Moderate response | 23.6
  Week 8: No response: number analyzed (Participants) | 93
  Week 8: No response | 65.6
  Week 12: Good response: number analyzed (Participants) | 87
  Week 12: Good response | 9.2
  Week 12: Moderate response: number analyzed (Participants) | 87
  Week 12: Moderate response | 20.7
  Week 12: No response: number analyzed (Participants) | 87
  Week 12: No response | 70.1
  Week 16: Good response: number analyzed (Participants) | 85
  Week 16: Good response | 5.9
  Week 16: Moderate response: number analyzed (Participants) | 85
  Week 16: Moderate response | 15.3
  Week 16: No response: number analyzed (Participants) | 85
  Week 16: No response | 78.8
  Week 20: Good response: number analyzed (Participants) | 82
  Week 20: Good response | 6.1
  Week 20: Moderate response: number analyzed (Participants) | 82
  Week 20: Moderate response | 26.8
  Week 20: No response: number analyzed (Participants) | 82
  Week 20: No response | 67.1
  Week 24: Good response: number analyzed (Participants) | 80
  Week 24: Good response | 6.2
  Week 24: Moderate response: number analyzed (Participants) | 80
  Week 24: Moderate response | 21.2
  Week 24: No response: number analyzed (Participants) | 80
  Week 24: No response | 72.6
  Week 28: Good response: number analyzed (Participants) | 79
  Week 28: Good response | 6.3
  Week 28: Moderate response: number analyzed (Participants) | 79
  Week 28: Moderate response | 11.4
  Week 28: No response: number analyzed (Participants) | 79
  Week 28: No response | 82.3
  Week 32: Good response: number analyzed (Participants) | 74
  Week 32: Good response | 0
  Week 32: Moderate response: number analyzed (Participants) | 74
  Week 32: Moderate response | 18.9
  Week 32: No response: number analyzed (Participants) | 74
  Week 32: No response | 81.1
  Week 36: Good response: number analyzed (Participants) | 74
  Week 36: Good response | 1.3
  Week 36: Moderate response: number analyzed (Participants) | 74
  Week 36: Moderate response | 14.9
  Week 36: No response: number analyzed (Participants) | 74
  Week 36: No response | 83.8
  Week 40: Good response: number analyzed (Participants) | 74
  Week 40: Good response | 5.4
  Week 40: Moderate response: number analyzed (Participants) | 74
  Week 40: Moderate response | 17.6
  Week 40: No response: number analyzed (Participants) | 74
  Week 40: No response | 77
  Week 44: Good response: number analyzed (Participants) | 72
  Week 44: Good response | 2.8
  Week 44: Moderate response: number analyzed (Participants) | 72
  Week 44: Moderate response | 13.9
  Week 44: No response: number analyzed (Participants) | 72
  Week 44: No response | 83.3
  Week 48: Good response: number analyzed (Participants) | 71
  Week 48: Good response | 5.7
  Week 48: Moderate response: number analyzed (Participants) | 71
  Week 48: Moderate response | 11.4
  Week 48: No response: number analyzed (Participants) | 71
  Week 48: No response | 82.9
  Week 52: Good response: number analyzed (Participants) | 67
  Week 52: Good response | 94
  Week 52: Moderate response: number analyzed (Participants) | 67
  Week 52: Moderate response | 6
  Week 52: No response: number analyzed (Participants) | 67
  Week 52: No response | 0

7. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score up to Week 52
Description: SDAI is an index for measuring disease activity. SDAI is the numerical sum of five outcome parameters: TJC28 and SJC28, PGA and physician global assessment of disease activity assessed on VAS (0 centimeter [cm]-10 cm); 0 cm= no disease activity and 10 cm= worst disease activity, and CRP (in milligrams per deciliter [mg/dL]). SDAI total score ranges from 0 to 86, with higher scores indicating increased (or severe) disease activity. SDAI score </=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
units on a scale
  Change at Week 2 | -3.41 [-7.17 to 0.12]
  Change at Week 4: number analyzed (Participants) | 95
  Change at Week 4 | -6.54 [-10.26 to -2.97]
  Change at Week 8: number analyzed (Participants) | 93
  Change at Week 8 | -8.72 [-12.89 to -5.18]
  Change at Week 12: number analyzed (Participants) | 87
  Change at Week 12 | -11.07 [-14.74 to -8.04]
  Change at Week 16: number analyzed (Participants) | 85
  Change at Week 16 | -13.47 [-17.00 to -10.60]
  Change at Week 20: number analyzed (Participants) | 82
  Change at Week 20 | -13.88 [-17.42 to -10.94]
  Change at Week 24: number analyzed (Participants) | 80
  Change at Week 24 | -14.08 [-17.72 to -11.25]
  Change at Week 28: number analyzed (Participants) | 79
  Change at Week 28 | -15.37 [-18.87 to -12.41]
  Change at Week 32: number analyzed (Participants) | 74
  Change at Week 32 | -16.09 [-19.63 to -13.07]
  Change at Week 36: number analyzed (Participants) | 74
  Change at Week 36 | -15.61 [-19.14 to -12.58]
  Change at Week 40: number analyzed (Participants) | 74
  Change at Week 40 | -14.86 [-18.66 to -11.84]
  Change at Week 44: number analyzed (Participants) | 71
  Change at Week 44 | -16.31 [-20.06 to -13.24]
  Change at Week 48: number analyzed (Participants) | 70
  Change at Week 48 | -16.47 [-20.13 to -13.45]
  Change at Week 52: number analyzed (Participants) | 67
  Change at Week 52 | -17.35 [-21.01 to -14.16]

8. Secondary Outcome: Change From Baseline in TJC28 up to Week 52
Description: 28 joints were assessed for tenderness and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 28. A negative change from baseline indicated improvement.
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
tender joints
  Change at Week 2 | -1.30 [-3.18 to 0.56]
  Change at Week 4: number analyzed (Participants) | 95
  Change at Week 4 | -3.26 [-5.09 to -1.42]
  Change at Week 8: number analyzed (Participants) | 93
  Change at Week 8 | -4.97 [-6.69 to -3.25]
  Change at Week 12: number analyzed (Participants) | 87
  Change at Week 12 | -5.82 [-7.55 to -4.09]
  Change at Week 16: number analyzed (Participants) | 85
  Change at Week 16 | -6.39 [-8.08 to -4.70]
  Change at Week 20: number analyzed (Participants) | 82
  Change at Week 20 | -7.03 [-8.67 to -5.38]
  Change at Week 24: number analyzed (Participants) | 80
  Change at Week 24 | -7.72 [-9.34 to -6.09]
  Change at Week 28: number analyzed (Participants) | 79
  Change at Week 28 | -7.91 [-9.51 to -6.31]
  Change at Week 32: number analyzed (Participants) | 74
  Change at Week 32 | -8.38 [-10.00 to -6.77]
  Change at Week 36: number analyzed (Participants) | 74
  Change at Week 36 | -8.28 [-9.86 to -6.66]
  Change at Week 40: number analyzed (Participants) | 74
  Change at Week 40 | -8.22 [-9.84 to -6.59]
  Change at Week 44: number analyzed (Participants) | 71
  Change at Week 44 | -8.63 [-10.25 to -7.01]
  Change at Week 48: number analyzed (Participants) | 70
  Change at Week 48 | -8.26 [-9.97 to -6.54]
  Change at Week 52: number analyzed (Participants) | 67
  Change at Week 52 | -8.75 [-10.41 to -7.09]

9. Secondary Outcome: Change From Baseline in SJC28 up to Week 52
Description: 28 joints were assessed for swelling and joints were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 28. A negative change from baseline indicated improvement.
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 96
swollen joints
  Change at Week 2 | -1.82 [-3.51 to -0.13]
  Change at Week 4: number analyzed (Participants) | 95
  Change at Week 4 | -3.08 [-4.70 to -1.46]
  Change at Week 8: number analyzed (Participants) | 93
  Change at Week 8 | -4.71 [-6.20 to -3.21]
  Change at Week 12: number analyzed (Participants) | 87
  Change at Week 12 | -5.24 [-6.68 to -3.79]
  Change at Week 16: number analyzed (Participants) | 85
  Change at Week 16 | -5.79 [-7.27 to -4.31]
  Change at Week 20: number analyzed (Participants) | 82
  Change at Week 20 | -6.06 [-7.55 to -4.57]
  Change at Week 24: number analyzed (Participants) | 80
  Change at Week 24 | -6.60 [-8.03 to -5.18]
  Change at Week 28: number analyzed (Participants) | 79
  Change at Week 28 | -6.65 [-8.09 to -5.21]
  Change at Week 32: number analyzed (Participants) | 74
  Change at Week 32 | -6.73 [-8.19 to -5.27]
  Change at Week 36: number analyzed (Participants) | 74
  Change at Week 36 | -6.76 [-8.22 to -5.28]
  Change at Week 40: number analyzed (Participants) | 74
  Change at Week 40 | -6.91 [-8.37 to -5.44]
  Change at Week 44: number analyzed (Participants) | 71
  Change at Week 44 | -6.82 [-8.31 to -5.33]
  Change at Week 48: number analyzed (Participants) | 70
  Change at Week 48 | -6.63 [-8.15 to -5.10]
  Change at Week 52: number analyzed (Participants) | 67
  Change at Week 52 | -6.98 [-8.52 to -5.44]

10. Secondary Outcome: Percentage of Participants With Corticosteroid Dose Reduction or Discontinuation
Time Frame: From Baseline up to Week 52
Population: Full analysis set. Overall number of participants analyzed = participants who used corticosteroids during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 37
percentage of participants | 48.6

11. Secondary Outcome: Number of Participants by Reasons (Categories) for Corticosteroid Dose Reduction or Discontinuation
Description: Reasons for corticosteroid dose reduction included: Safety Reasons (including elevated liver function test results, respiratory infections, infections and infestations, gastrointestinal disorders etc.); Other Reasons (disease remission, improvement etc.); and Unknown Reasons (including no reason). Number of participants by reasons (Safety, Other, Unknown) for corticosteroid dose reduction or discontinuation were reported.
Time Frame: From Baseline up to Week 52
Population: Full analysis set. Overall number of participants analyzed = participants with corticosteroid dose reduction/discontinuation.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 18
participants
  Safety | 6
  Other | 10
  Unknown | 2

12. Secondary Outcome: Number of Participants With Anti-Tocilizumab Antibodies (ATA)
Description: All samples were tested using a screening assay and, if positive, by a confirmation assay to determine specificity and a neutralizing assay to test for the ability to inhibit the activity of tocilizumab. Number of participants with a positive assay result for screening assay (ATA - Screen), confirmatory assay (ATA - Confirmatory), and neutralizing assay (ATA - Neutralizing) was reported separately.
Time Frame: Baseline (Week 1), Weeks 12, 24, 36, 52, and 8 weeks after Week 52 dose (Week 60)
Population: Full analysis set. Here, Number analyzed = number of participants analyzed for this outcome measure at specified timepoint.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
participants
  Week 1: ATA - Screen | 7
  Week 1: ATA - Confirmatory | 4
  Week 1: ATA - Neutralizing | 0
  Week 12: ATA - Screen: number analyzed (Participants) | 87
  Week 12: ATA - Screen | 3
  Week 12: ATA - Confirmatory: number analyzed (Participants) | 87
  Week 12: ATA - Confirmatory | 0
  Week 12: ATA - Neutralizing: number analyzed (Participants) | 87
  Week 12: ATA - Neutralizing | 0
  Week 24: ATA - Screen: number analyzed (Participants) | 78
  Week 24: ATA - Screen | 3
  Week 24: ATA - Confirmatory: number analyzed (Participants) | 78
  Week 24: ATA - Confirmatory | 1
  Week 24: ATA - Neutralizing: number analyzed (Participants) | 78
  Week 24: ATA - Neutralizing | 1
  Week 36: ATA - Screen: number analyzed (Participants) | 73
  Week 36: ATA - Screen | 2
  Week 36: ATA - Confirmatory: number analyzed (Participants) | 73
  Week 36: ATA - Confirmatory | 0
  Week 36: ATA - Neutralizing: number analyzed (Participants) | 73
  Week 36: ATA - Neutralizing | 0
  Week 52: ATA - Screen: number analyzed (Participants) | 67
  Week 52: ATA - Screen | 2
  Week 52: ATA - Confirmatory: number analyzed (Participants) | 67
  Week 52: ATA - Confirmatory | 0
  Week 52: ATA - Neutralizing: number analyzed (Participants) | 67
  Week 52: ATA - Neutralizing | 0
  Week 60: ATA - Screen: number analyzed (Participants) | 41
  Week 60: ATA - Screen | 1
  Week 60: ATA - Confirmatory: number analyzed (Participants) | 41
  Week 60: ATA - Confirmatory | 1
  Week 60: ATA - Neutralizing: number analyzed (Participants) | 41
  Week 60: ATA - Neutralizing | 0

13. Secondary Outcome: Soluble Interleukin-6 Receptor (sIL-6R) Levels
Time Frame: Baseline (Week 1), Weeks 12, 24, 36, 52, and 8 weeks after Week 52 dose (Week 60)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
nanograms per milliliter (ng/mL)
  Week 1 | 39450 (10740)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 553.43 (120.36)
  Week 24: number analyzed (Participants) | 78
  Week 24 | 572.03 (136.68)
  Week 36: number analyzed (Participants) | 73
  Week 36 | 570.78 (139.16)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 537.73 (152.55)
  Week 60: number analyzed (Participants) | 41
  Week 60 | 42850 (13800)

14. Secondary Outcome: Tocilizumab Serum Levels
Time Frame: Baseline (Week 1), Weeks 12, 24, 36, 52, and 8 weeks after Week 52 dose (Week 60)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgrms per milliliter (mcg/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
microgrms per milliliter (mcg/mL)
  Week 1 | 0.38 (0.17)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 41.98 (25.04)
  Week 24: number analyzed (Participants) | 78
  Week 24 | 44.67 (28.83)
  Week 36: number analyzed (Participants) | 73
  Week 36 | 47.90 (28.29)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 45.37 (28.13)
  Week 60: number analyzed (Participants) | 41
  Week 60 | 6.46 (4.28)

15. Secondary Outcome: PGA, Using VAS Score
Description: PGA was assessed on a 0 to 100 mm horizontal VAS. The extreme left end of the line = 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end = 100 mm, and was described as "maximum disease activity" (maximum arthritis disease activity). Higher values correspond to worst state of participant (high disease activity).
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
mm
  Week 1 | 28.26 (20.25)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 27.57 (20.08)
  Week 4: number analyzed (Participants) | 95
  Week 4 | 28.36 (19.37)
  Week 8: number analyzed (Participants) | 93
  Week 8 | 32.28 (22.09)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 28.73 (23.01)
  Week 16: number analyzed (Participants) | 85
  Week 16 | 24.40 (19.02)
  Week 20: number analyzed (Participants) | 82
  Week 20 | 28.15 (20.22)
  Week 24: number analyzed (Participants) | 80
  Week 24 | 32.63 (23.44)
  Week 28: number analyzed (Participants) | 79
  Week 28 | 26.02 (18.79)
  Week 32: number analyzed (Participants) | 74
  Week 32 | 27.08 (20.98)
  Week 36: number analyzed (Participants) | 74
  Week 36 | 30.79 (22.37)
  Week 40: number analyzed (Participants) | 74
  Week 40 | 30.50 (21.93)
  Week 44: number analyzed (Participants) | 71
  Week 44 | 25.79 (16.33)
  Week 48: number analyzed (Participants) | 70
  Week 48 | 23.86 (19.11)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 23.08 (17.08)

16. Secondary Outcome: Patient Assessment of Pain, Using VAS Score
Description: The participant's level of pain was assessed on a 0 to 100 mm horizontal VAS. The extreme left end of the line = 0 mm, and was described as "no pain" and the extreme right end = 100 mm, and was described as "unbearable pain". Higher values correspond to worst state of participant (higher level of pain).
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
mm
  Week 1 | 46.40 (27.43)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 52.04 (24.46)
  Week 4: number analyzed (Participants) | 95
  Week 4 | 49.87 (23.35)
  Week 8: number analyzed (Participants) | 93
  Week 8 | 42.72 (23.20)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 37.21 (21.29)
  Week 16: number analyzed (Participants) | 85
  Week 16 | 34.24 (22.49)
  Week 20: number analyzed (Participants) | 82
  Week 20 | 31.00 (19.42)
  Week 24: number analyzed (Participants) | 80
  Week 24 | 29.57 (19.66)
  Week 28: number analyzed (Participants) | 79
  Week 28 | 29.63 (19.07)
  Week 32: number analyzed (Participants) | 74
  Week 32 | 25.50 (17.95)
  Week 36: number analyzed (Participants) | 74
  Week 36 | 26.78 (22.13)
  Week 40: number analyzed (Participants) | 74
  Week 40 | 27.50 (21.93)
  Week 44: number analyzed (Participants) | 71
  Week 44 | 26.88 (19.96)
  Week 48: number analyzed (Participants) | 70
  Week 48 | 23.61 (18.63)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 23.98 (20.19)

17. Secondary Outcome: HAQ-DI Score
Description: The Stanford HAQ-DI is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Responses in each component set were scored from 0 (without any difficulty) to 3 (unable to do). The highest score recorded for any question in a category determines the score for the category, unless aids, devices, or help from another person was required. The HAQ-DI score was calculated as the sum of the category scores divided by the number of categories scored, giving a possible range of scores from 0 to 3. Scores of 0 to 1 are generally considered to represent "mild to moderate difficulty", 1 to 2 as "moderate to severe disability", and 2 to 3 as "severe to very severe disability".
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
units on a scale
  Week 1 | 1.31 (0.66)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 1.22 (0.64)
  Week 4: number analyzed (Participants) | 95
  Week 4 | 1.09 (0.66)
  Week 8: number analyzed (Participants) | 93
  Week 8 | 0.91 (0.66)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 0.82 (0.58)
  Week 16: number analyzed (Participants) | 85
  Week 16 | 0.72 (0.59)
  Week 20: number analyzed (Participants) | 82
  Week 20 | 0.68 (0.56)
  Week 24: number analyzed (Participants) | 80
  Week 24 | 0.66 (0.55)
  Week 28: number analyzed (Participants) | 79
  Week 28 | 0.66 (0.57)
  Week 32: number analyzed (Participants) | 74
  Week 32 | 0.59 (0.58)
  Week 36: number analyzed (Participants) | 74
  Week 36 | 0.63 (0.58)
  Week 40: number analyzed (Participants) | 74
  Week 40 | 0.60 (0.59)
  Week 44: number analyzed (Participants) | 71
  Week 44 | 0.59 (0.61)
  Week 48: number analyzed (Participants) | 70
  Week 48 | 0.56 (0.59)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 0.54 (0.60)

18. Secondary Outcome: Percentage of Participants Who Received All Planned Study Medication (Compliance)
Description: Compliance (in terms of percentage of participants who received all planned study medication) was assessed on the basis of participant diary cards and return records.
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
percentage of participants
  Week 1 | 66
  Week 2: number analyzed (Participants) | 96
  Week 2 | 97.9
  Week 4: number analyzed (Participants) | 95
  Week 4 | 100
  Week 8: number analyzed (Participants) | 93
  Week 8 | 100
  Week 12: number analyzed (Participants) | 87
  Week 12 | 98.9
  Week 16: number analyzed (Participants) | 85
  Week 16 | 97.6
  Week 20: number analyzed (Participants) | 82
  Week 20 | 98.8
  Week 24: number analyzed (Participants) | 80
  Week 24 | 100
  Week 28: number analyzed (Participants) | 79
  Week 28 | 100
  Week 32: number analyzed (Participants) | 74
  Week 32 | 100
  Week 36: number analyzed (Participants) | 74
  Week 36 | 100
  Week 40: number analyzed (Participants) | 74
  Week 40 | 100
  Week 44: number analyzed (Participants) | 71
  Week 44 | 100
  Week 48: number analyzed (Participants) | 70
  Week 48 | 100
  Week 52: number analyzed (Participants) | 67
  Week 52 | 100

19. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score
Description: FACIT-Fatigue total score is sum of FACIT-General subscale score and FACIT-Fatigue (additional concerns) subscale score. FACT-General consists of 27 questions grouped in 4 domains of general health-related quality of life: physical well-being, social/family well-being, emotional well-being, and functional well-being; each item ranges from 0 (not at all) to 4 (very much). FACT-General score ranges between 0-108. FACIT-Fatigue subscale is a 13-item questionnaire that evaluates self-reported fatigue and its impact upon daily activities. Each item ranges from 0 (Not at all) to 4 (Very much). For all items, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue subscale score for a total possible score of 0 (worse score) to 52 (better score). FACIT-Fatigue total score (FACT-G plus FACT-F subscale scores) ranges from 0 (better score) to 160 (worse score).
Time Frame: Baseline (Week 1), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
units on a scale
  Week 1 | 89.68 (24.32)
  Week 2: number analyzed (Participants) | 96
  Week 2 | 91.83 (22.91)
  Week 4: number analyzed (Participants) | 95
  Week 4 | 100.38 (24.36)
  Week 8: number analyzed (Participants) | 93
  Week 8 | 103.16 (26.28)
  Week 12: number analyzed (Participants) | 87
  Week 12 | 106.39 (24.74)
  Week 16: number analyzed (Participants) | 85
  Week 16 | 110.17 (24.96)
  Week 20: number analyzed (Participants) | 82
  Week 20 | 112.60 (25.50)
  Week 24: number analyzed (Participants) | 80
  Week 24 | 114.21 (25.23)
  Week 28: number analyzed (Participants) | 79
  Week 28 | 114.85 (26.95)
  Week 32: number analyzed (Participants) | 74
  Week 32 | 117.01 (26.00)
  Week 36: number analyzed (Participants) | 74
  Week 36 | 116.50 (26.17)
  Week 40: number analyzed (Participants) | 74
  Week 40 | 116.59 (26.20)
  Week 44: number analyzed (Participants) | 71
  Week 44 | 119.67 (26.64)
  Week 48: number analyzed (Participants) | 70
  Week 48 | 119.83 (26.51)
  Week 52: number analyzed (Participants) | 67
  Week 52 | 121.82 (25.34)

ADVERSE EVENTS:
Time Frame: From Baseline up to end of study (Week 60)
Description: Safety population included all participants who received at least one dose of SC tocilizumab. Adverse events were reported separately for the participants who received tocilizumab monotherapy and tocilizumab in combination with methotrexate or other non-biologic DMARDs.
Groups:
- Tocilizumab Monotherapy: Participants received tocilizumab 162 mg SC injection QW as monotherapy during the treatment period of 52 weeks.
- Tocilizumab + Methotrexate or Other Non-Biologic DMARDs: Participants received tocilizumab 162 mg SC injection QW in combination with methotrexate or other non-biologic DMARDs during the treatment period of 52 weeks.
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + Methotrexate or Other Non-Biologic DMARDs
Serious Adverse Events (participants affected / at risk) | 2/31 | 5/66
Other Adverse Events (participants affected / at risk) | 19/31 | 38/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=31) | Tocilizumab + Methotrexate or Other Non-Biologic DMARDs (N=66)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=31) | Tocilizumab + Methotrexate or Other Non-Biologic DMARDs (N=66)
Leukopenia (Blood and lymphatic system disorders) | 4 | 8
Lymphopenia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 6 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 4 | 0
Injection site erythema (General disorders) | 1 | 5
Oedema peripheral (General disorders) | 2 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 6
Bronchitis (Infections and infestations) | 3 | 5
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 2 | 5
Contusion (Injury, poisoning and procedural complications) | 3 | 2
Alanine aminotransferase increased (Investigations) | 9 | 13
Aspartate aminotransferase increased (Investigations) | 8 | 9
Blood glucose increased (Investigations) | 2 | 3
Blood triglycerides increased (Investigations) | 3 | 3
Blood urea increased (Investigations) | 1 | 3
Blood uric acid increased (Investigations) | 3 | 1
Hepatic enzyme increased (Investigations) | 1 | 5
White blood cell count decreased (Investigations) | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Hypertension (Vascular disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Injection site pruritus (General disorders) | 2 | 1
Neutrophil count decreased (Investigations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.